CLINICAL TRIAL: NCT05210634
Title: A Two-Phase, Randomized, Double-Blind, PlaceboControlled Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of CHI-915 in Healthy Participants
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of CHI-915 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Canopy Growth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 710022US1312
Record Dates: First submitted 2021-12-31; First posted 2022-01-27 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: The is a two-phase, within participant crossover study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Phase 1 will follow a single-ascending dose design in 3 participants. This portion of the study will be unblinded. Phase 2 will follow a within-participant crossover design in 15 participants. Participants will be randomized to a dosing order. Phase 2 is double-blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: Placebo (Placebo Comparator): Single oral administration of 4 ml of Placebo MCT oil
  Interventions: Dietary Supplement: THCv
- Group 2: 12.5 mg THCv (CHI-915) (Active Comparator): Single oral administration of 12.5 mg THCv in MCT oil
  Interventions: Dietary Supplement: THCv
- Group 3: 25 mg THCv (CHI-915) (Active Comparator): Single oral administration of 25 mg THCv in MCT oil
  Interventions: Dietary Supplement: THCv
- Group 4: 50 mg THCv (CHI-915) (Active Comparator): Single oral administration of 50 mg THCv in MCT oil
  Interventions: Dietary Supplement: THCv
- Group 5: 100 mg THCv (CHI-915) (Active Comparator): Single oral administration of 100 mg THCv in MCT oil
  Interventions: Dietary Supplement: THCv
- Group 6: 200 mg THCv (CHI-915) (Active Comparator): Single oral administration of 200 mg THCv in MCT oil
  Interventions: Dietary Supplement: THCv

INTERVENTIONS:
Dietary Supplement: THCv — THCv in MCT oil

SUMMARY:
This is a two-phase, randomized, double-blind, placebo-controlled, within-participant crossover study to assess the safety, tolerability, PK, and PD of five oral doses of CHI-915 versus placebo in healthy adult participants ages 18-55 years.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult aged 18-55 years (inclusive) at the time of screening.
2. Has a body mass index between 18 and 30 kg/m2.
3. Is judged by the Investigator to be in generally good health at screening based on the results of a medical history, physical examination, 12-lead ECG, and clinical laboratory test results. Laboratory results outside of the reference range deemed to be acceptable will be documented as not clinically significant at the discretion of the Investigator.
4. For women of childbearing potential, has a negative serum pregnancy test (β-human chorionic gonadotropin [hCG]) at the Screening Visit and a negative urine pregnancy test at intake to the research facility.
5. Must be adequately informed of the nature and risks of the study and give written informed consent prior to screening.
6. Is, in the Investigator's opinion, reliable, able, and willing to comply with all protocol requirements and procedures (including scheduled visits).

Exclusion Criteria:

1. Women who are pregnant, lactating, breastfeeding, or planning a pregnancy.
2. Women of childbearing potential, or men who are sexually active with a woman of childbearing potential, who are unwilling or unable to use an acceptable method of contraception (abstinence or the use of a highly effective method of contraception, including hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom, vasectomy, or intrauterine device) from at least 21 days prior to the first dose of study medication until 28 days after the last dose of study medication. Participants with same sex partners or who maintain abstinence do not require contraception.
3. Person has history of diagnosis related to hepatic function and/or significantly impaired hepatic function (alanine aminotransferase [ALT] >3x upper limit of normal [ULN] or total bilirubin [TBL] >2 x ULN) OR the ALT or aspartate aminotransferase (AST) >2 x ULN and TBL >2 x ULN (or international normalized ratio [INR] >1.5).
4. Has a history of epilepsy.
5. Has used tobacco/nicotine-containing products on more than 10 occasions within 30 days of dosing with study IP or during the study.
6. Has used any prescription drugs or herbal supplements (except hormonal contraception) within 30 days prior to receiving the first dose of IP, unless approved by the Investigator and stable for at least 30 days prior to the first dose of IP through the final study visit.
7. Use of any over-the-counter drugs, vitamins, or supplements within 24 hours prior to dosing with the IP.
8. Has or has previously had a positive result for the presence of Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibodies (HCVAb), or human immunodeficiency virus (HIV) antibodies.
9. Has a positive breath, urine, or serum test for ethanol or a positive urine screen for cocaine, THC, barbiturates, amphetamines, methamphetamines, benzodiazepines, methylenedioxymethamphetamine, phencyclidine, methadone, or opiates at the Screening Visit or prior to IP administration.
10. Any clinically significant condition or abnormal finding at the Screening Visit that would, in the opinion of the Investigator, preclude study participation or interfere with evaluation of the IP.
11. Has a history of a known significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to any compound or chemical class related to cannabis, including phytocannabinoids and cannabinoid analogues, or excipients utilized within the IP.
12. Has taken grapefruit products and/or Seville oranges within the 7 days prior to dosing with study medication or during the study.
13. Is taking a prohibited medication or supplement including warfarin, clobazam, valproic acid, phenobarbital, mTOR inhibitors, oral tacrolimus, and St. John's Wort within 30 days prior to receiving the first dose of IP or during the study.
14. Has used cannabis, synthetic cannabinoid, or cannabinoid analogues (e.g., dronabinol, nabilone), hemp products, synthetic cannabinoid receptor agonists (e.g., spice, K2), or any cannabidiol (CBD) or THC-containing product (e.g., Sativex, Epidiolex) within 4 weeks of the Screening Visit or during the study and has used cannabis on more than 25 occasions in the last 12 months.
15. Meets criteria for past-year Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)-defined psychiatric disorder, or moderate to severe substance use disorder.
16. Has a lifetime history of psychosis or schizophrenia or a first-degree relative experiencing psychosis or schizophrenia.
17. Endorses current suicidal intent as indexed by endorsement of questions #4 or #5 on the Columbia-Suicide Severity Rating Scale (C-SSRS).
18. Has suspected or confirmed cardiovascular disease.
19. Has participated in any investigational product or device study within 30 days prior to receiving the first dose of IP or is scheduled to participate in another investigational product or device study during the course of this study.
20. Demonstrates behavior indicating unreliability or inability to comply with the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Incidence, type and severity of AEs/SAEs | Day 1
  Incidence, type and severity of AEs/SAEs
Incidence, type and severity of AEs/SAEs | Day 8
  Incidence, type and severity of AEs/SAEs
Incidence, type and severity of AEs/SAEs | Day 15
  Incidence, type and severity of AEs/SAEs
Incidence, type and severity of AEs/SAEs | Day 22
  Incidence, type and severity of AEs/SAEs
Incidence, type and severity of AEs/SAEs | Day 29
  Incidence, type and severity of AEs/SAEs
Incidence, type and severity of AEs/SAEs | Day 36
  Incidence, type and severity of AEs/SAEs
Change in blood pressure | Day 1
  Change in systolic and diastolic blood pressure measured in mmHg
Change in heart rate | Day 1
  Change in heart rate measured in beats per minute
Change in respiratory rate | Day 1
  Change in respiratory rate measured in breaths per minute
Change in body temperature | Day 1
  Change in body temperature measured in degrees Celsius
Change in blood pressure | Day 8
  Change in systolic and diastolic blood pressure measured in mmHg
Change in heart rate | Day 8
  Change in heart rate measured in beats per minute
Change in respiratory rate | Day 8
  Change in respiratory rate measured in breaths per minute
Change in body temperature | Day 8
  Change in body temperature measured in degrees Celsius
Change in blood pressure | Day 15
  Change in systolic and diastolic blood pressure measured in mmHg
Change in respiratory rate | Day 15
  Change in respiratory rate measured in breaths per minute
Change in heart rate | Day 15
  Change in heart rate measured in beats per minute
Change in body temperature | Day 15
  Change in body temperature measured in degrees Celsius
Change in blood pressure | Day 22
  Change in systolic and diastolic blood pressure measured in mmHg
Change in respiratory rate | Day 22
  Change in respiratory rate measured in breaths per minute
Change in heart rate | Day 22
  Change in heart rate measured in beats per minute
Change in body temperature | Day 22
  Change in body temperature measured in degrees Celsius
Change in blood pressure | Day 29
  Change in systolic and diastolic blood pressure measured in mmHg
Change in heart rate | Day 29
  Change in heart rate measured in beats per minute
Change in respiratory rate | Day 29
  Change in respiratory rate measured in breaths per minute
Change in body temperature | Day 29
  Change in body temperature measured in degrees Celsius
Change in blood pressure | Day 36
  Change in systolic and diastolic blood pressure measured in mmHg
Change in heart rate | Day 36
  Change in heart rate measured in beats per minute
Change in respiratory rate | Day 36
  Change in respiratory rate measured in breaths per minute
Change in body temperature | Day 36
  Change in body temperature measured in degrees Celsius
Change in ECG results | Day 1
  Change in ECG results. Results summarized as Normal, Abnormal not clinically significant, and Abnormal clinically significant
Change in ECG results | Day 8
  Change in ECG results. Results summarized as Normal, Abnormal not clinically significant, and Abnormal clinically significant
Change in ECG results | Day 15
  Change in ECG results. Results summarized as Normal, Abnormal not clinically significant, and Abnormal clinically significant
Change in ECG results | Day 22
  Change in ECG results. Results summarized as Normal, Abnormal not clinically significant, and Abnormal clinically significant
Change in ECG results | Day 29
  Change in ECG results. Results summarized as Normal, Abnormal not clinically significant, and Abnormal clinically significant
Change in ECG results | Day 36
  Change in ECG results. Results summarized as Normal, Abnormal not clinically significant, and Abnormal clinically significant

SECONDARY OUTCOMES:
Maximum effect for the item "energetic" on the DEQ | Day 1
  Maximum effect for the item "energetic" on the Drug Effects Questionnaire. Scale from 0-100 where higher scores indicate more "energetic"
Maximum effect for the item "energetic" on the DEQ | Day 8
  Maximum effect for the item "energetic" on the Drug Effects Questionnaire. Scale from 0-100 where higher scores indicate more "energetic"
Maximum effect for the item "energetic" on the DEQ | Day 15
  Maximum effect for the item "energetic" on the Drug Effects Questionnaire. Scale from 0-100 where higher scores indicate more "energetic"
Maximum effect for the item "energetic" on the DEQ | Day 22
  Maximum effect for the item "energetic" on the Drug Effects Questionnaire. Scale from 0-100 where higher scores indicate more "energetic"
Maximum effect for the item "energetic" on the DEQ | Day 29
  Maximum effect for the item "energetic" on the Drug Effects Questionnaire. Scale from 0-100 where higher scores indicate more "energetic"
Maximum effect for the item "energetic" on the DEQ | Day 36
  Maximum effect for the item "energetic" on the Drug Effects Questionnaire. Scale from 0-100 where higher scores indicate more "energetic"
Sustained attention - maximum total time on the DVT | Day 1
  Sustained attention - maximum total time on the DVT
Sustained attention - maximum total time on the DVT | Day 8
  Sustained attention - maximum total time on the DVT
Sustained attention - maximum total time on the DVT | Day 15
  Sustained attention - maximum total time on the DVT
Sustained attention - maximum total time on the DVT | Day 22
  Sustained attention - maximum total time on the DVT
Sustained attention - maximum total time on the DVT | Day 29
  Sustained attention - maximum total time on the DVT
Sustained attention - maximum total time on the DVT | Day 36
  Sustained attention - maximum total time on the DVT
Pharmacokinetic profile of THCv | Day 1
  Pharmacokinetic profile of THCv measured by maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 8
  Pharmacokinetic profile of THCv measured by maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 15
  Pharmacokinetic profile of THCv measured by maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 22
  Pharmacokinetic profile of THCv measured by maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 29
  Pharmacokinetic profile of THCv measured by maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 36
  Pharmacokinetic profile of THCv measured by maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 1
  Pharmacokinetic profile of THCv measured by time to maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 8
  Pharmacokinetic profile of THCv measured by time to maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 15
  Pharmacokinetic profile of THCv measured by time to maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 22
  Pharmacokinetic profile of THCv measured by time to maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 29
  Pharmacokinetic profile of THCv measured by time to maximum observed plasma concentration
Pharmacokinetic profile of THCv | Day 36
  Pharmacokinetic profile of THCv measured by time to maximum observed plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Sempio C, Campos-Palomino J, Klawitter J, Peters EN, MacNair L, Haghdoost M, Bonn-Miller MO, Harrison A, Babalonis S, Christians U, Klawitter J. Pharmacokinetics of Oral Cannabinoid Delta8-Tetrahydrocannabivarin and Its Main Metabolites in Healthy Participants. Pharmaceuticals (Basel). 2024 Nov 27;17(12):1603. doi: 10.3390/ph17121603. PMID 39770444
- [Derived] Peters EN, MacNair L, Harrison A, Feldner MT, Eglit GML, Babalonis S, Turcotte C, Bonn-Miller MO. A Two-Phase, Dose-Ranging, Placebo-Controlled Study of the Safety and Preliminary Test of Acute Effects of Oral Delta8-Tetrahydrocannabivarin in Healthy Participants. Cannabis Cannabinoid Res. 2023 Sep;8(S1):S71-S82. doi: 10.1089/can.2023.0038. PMID 37721990